CLINICAL TRIAL: NCT03693664
Title: Validity and Reliability of the 6-Minute Pegboard and Ring Test Unsupported Arm Function Exercise Test in Controlled and Partially Controlled Asthma Patients
Brief Title: 6-Minute Pegboard and Ring Test Unsupported Arm Function Exercise Test in Asthma Patients
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, principal investigator, Hacettepe University
Other Study IDs: GO 18206/24
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Asthma
Keywords: Asthma; Daily Living Activities; 6 Minute Pegboard and Ring Test
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Exercise intolerance is one of the most problems in chronic obstructive pulmonary disease (COPD) and occurs not only in performing lower body tasks but also in performing arm activities. During arm exercise, auxiliary respiratory muscles are used for arm duty and cannot contribute to breathing. This increases the respiratory load of the diaphragm, which is mechanically disadvantageous, and results in thoracoabdominal synchronization disorder and severe dyspnea. Although the relationship between activity limitation and quality of life is clear in patients with exertional activity, the literature on physical activity is insufficient. Exercise and physical activity can also and exercise-related respiratory symptoms are known to have adverse effects on daily living activities (ADLs). There is no gold standard for objective assessment of activity limitation and exertional dyspnea in patients with asthma. Therefore, the results obtained by evaluating the validity and reliability of the 6PRT test in asthmatic patients in this study will increase the use of this test to test both arm endurance and arm exercise capacity in adult asthmatic patients, to estimate the effect on ADLs and to demonstrate the development obtained with pulmonary rehabilitation. .

DETAILED DESCRIPTION:
Objective: The aim of the study was to evaluate the validity and reliability of the six-minute pegboard and ring test in patients with controlled and partially controlled asthma.

* Demographic information: Name, age, diagnosis, occupation, body weight, height, The symptoms of the dominant and affected side, CV, family history, obstructive pulmonary diseases (dyspnoea, cough, incontinence frequency), clinical findings and respiratory function test parameters will be recorded.
* Assessment of Respiratory Muscle Strength: With intraoral pressure measurement instrument will be measured.
* Evaluation of Hand Grip Force: It will be measured by hand dynamometer.
* Unarmed Arm Exercise Capacity and Arm Function / Endurance Evaluation: '6 minute Pegboard and Ring Test-6PRT'. During the test, the patient is asked to sit in front of a perforated panel and to carry as many rings as possible for six minutes to the two upper holes using two hands at the same time. Participants are attached to the test by installing a few rings before the test. Standardized encouragement is given every minute during the test. The number of rings carried for 6 minutes constitutes the final score. Before and after the test, pulse oximetry and heart rate and oxygen saturation, modified Borg scale, dyspnea, general fatigue and arm fatigue are questioned. For the validity of the test, the test will be repeated in the same patient under the same conditions every one week.

  -Evaluation of Maximal Arm Exercise Capacity: With arm ergometer limited exercise test with maximal symptoms will be evaluated and used as a criterion for the reliability of 6PRT test.
* Daily life activities of dyspnea and breathlessness Evaluation of its Effect: The Modified Medical Research Council Scale will be evaluated with an objective measurement of 3 minutes breathing exercise test and London Chest Daily Living Activities Scale.
* Evaluation of Postural Awareness: The validity of the Turkish version developed by Shields, Mallory & Simon in 1989 will be evaluated by the Body Awareness Survey (VFA).
* Evaluation of Daily Living Activities: London Chest GYA Scale (25) and Milliken GYA Scale will be evaluated.
* Assessment of Quality of Life: Disease-specific Asthma Quality of Life Scale and Health Assessment Questionnaire.
* Asthma Control Assessment: Asthma Control Test will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* To have a controlled or partially controlled asthma diagnosis, Have not experienced acute exacerbation in the last 3 months, Being between 18-80 years of age, Volunteer for research, To be able to walk and cooperate.

Exclusion Criteria:

* To have a neurological disease or another clinical diagnosis that may affect cognitive status,
* To have musculoskeletal and neurological disease, symptomatic heart disease, previous lung surgery and malignant disease that may affect exercise performance.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Validity and reliability
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
6 minute Pegboard and Ring Test-6PRT | one year
  Total number of rings installed within six minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, Phd, Principal Investigator — Hacettepe University Physiotherapy and Rehabilitation
Locations (1):
- Hacettepe University, Ankara, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Calik-Kutukcu E, Tekerlek H, Bozdemir-Ozel C, Karaduz BN, Cakmak A, Inal-Ince D, Saglam M, Vardar-Yagli N, Sonbahar-Ulu H, Firat M, Arikan H, Kaya SB, Karakaya G. Validity and reliability of 6-minute pegboard and ring test in patients with asthma. J Asthma. 2022 Jul;59(7):1387-1395. doi: 10.1080/02770903.2021.1930040. Epub 2021 May 31. PMID 33985406